CLINICAL TRIAL: NCT00883714
Title: Exercise During the Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. Fernando Dimeo, Dept. of Sports Medicine, Charité Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EA4/030/09
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Fatigue; Allogeneic Stem Cell Transplantation
Keywords: Exercise; sport; Allogeneic blood stem cell transplantation; Blood stem cell transplantation; Fatigue; Cancer; Physical performance; Mood; Complications
MeSH Terms: conditions — Fatigue; Motor Activity; Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised exercise (Experimental)
  Interventions: Other: Supervised exercise
- Control group (Active Comparator)
  Interventions: Other: Exercise Instruction

INTERVENTIONS:
Other: Supervised exercise — The patients will carry out a daily exercise program consisting of walking on a treadmill for 30 minutes at an intensity of 80% of the maximum heart rate. The patients will be supervised by medical personnel.
  Arms: Supervised exercise
Other: Exercise Instruction — The patients will receive instructions about exercise and will have access to a bike ergometer to work out. However, they will not receive daily supervision or participate in a structured exercise program.
  Arms: Control group

SUMMARY:
The study will evaluate the effects of a structured endurance exercise program on the physical performance, the mood and the complications of patients with hematological malignancies undergoing a high-dose chemotherapy followed by an allogeneic peripheral blood stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Neoplastic malignancy
* Allogeneic peripheral stem cell transplantation
* Proficiency in German

Exclusion Criteria:

* Cardiorespiratory, metabolical, osteoarticular or immunological disorders which can be aggravated by exercise
* Pathological stress-ECG at admission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-04 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
VO2max | At recruitment and after 4 weeks

SECONDARY OUTCOMES:
Complications | 4 weeks
Mood | At recruitment and after 4 weeks
Requirement for blood and platelets transfusions | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dimeo, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Section Sports Medicine, Charité Universitätsmedizin Berlin, Hindenburgdamm 30, Berlin, State of Berlin, Germany